CLINICAL TRIAL: NCT06495138
Title: Daily Versus Intermittent Incremental Vestibulo-ocular Reflex Adaptation as a Novel Treatment for Dizziness in People With Multiple Sclerosis
Brief Title: Incremental Vestibulo-ocular Reflex Adaptation as a Novel Treatment for Dizziness in People With Multiple Sclerosis
Acronym: DIIVA-MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Colin R. Grove, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00007558; RG-2307-41945 (Other: National Multiple Sclerosis Society)
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis
Keywords: Treatment of multiple sclerosis; Incremental Vestibulo-ocular Reflex Adaptation; Dizziness in people with multiple sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Subjects will be block-randomized to one of two treatment groups. These groups will be stratified based on the region(s) of central nervous system involvement as determined by participants' Functional System Scores. During the six-week intervention phase, StableEyes will deliver either D-IVA-GSE or I-VA-GSE to participants based on their randomization results.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Daily Incremental Vestibulo-ocular Reflex Adaptation (D-IVA-GSE) (Experimental): The dosages of the D-IVA-GSE and I-IVA-GSE are based on the FITT principle of exercise prescription (frequency, intensity, time, and type). The D-IVA-GSE group will perform two, 15- minute GSE sessions (30-minutes total per day), seven days per week.
  Interventions: Device: StableEyes
- Intermittent incremental vestibulo-ocular Reflex Adaptation (I-IVA-GSE) (Experimental): The I-IVA-GSE group will perform two, 15-minute IVA-GSE sessions (30 minutes total), three days per week, with at least one day between each exercise day.
  Interventions: Device: StableEyes
- Helathy Control (No Intervention): The healthy control group will complete the same baseline assessments as the subjects in the Multiple Sclerosis (MS) group to serve as normative reference data.

INTERVENTIONS:
Device: StableEyes — Gaze stabilization exercises using the StableEyes device for the incremental vestibular-ocular reflex adaptation approach.
  The StableEyes device consists of a lightweight head unit with a 9-dimension inertial measurement unit and electrostatic micro-mirror that dynamically controls the 2-dimensional position of a 1-milliwatt red laser projected on a wall 1 meter in front of the subject. StableEyes is controlled via a lightweight control unit with a touchscreen interface tethered by cable to the head unit.
  Arms: Daily Incremental Vestibulo-ocular Reflex Adaptation (D-IVA-GSE); Intermittent incremental vestibulo-ocular Reflex Adaptation (I-IVA-GSE)

SUMMARY:
The study aims to study the effects of a novel treatment for vestibular symptoms in people with multiple sclerosis. The main objective is to determine whether daily personalized gaze stabilization training is more beneficial than intermittent gaze stability training in people with multiple sclerosis.

DETAILED DESCRIPTION:
People with multiple sclerosis (MS) often experience dizziness, caused by problems in how their brain processes balance signals. This dizziness can lead to difficulties keeping their eyes focused on a target while moving their head, known as gaze instability. This makes activities like walking or driving challenging and dangerous. Vestibular physical therapy, including gaze stabilization exercises, can help. The team developed StableEyes, a technology that improves gaze stability using a gradual approach to these exercises. In the studies, StableEyes significantly enhanced gaze stability in people with balance issues. Preliminary research in people with MS shows promising results, suggesting that tailored gaze stability exercises can further improve their vision stability. This method targets the vestibulo-ocular reflex (VOR), a critical reflex for maintaining clear vision during head movements. Improved VOR function can reduce dizziness and improve the quality of life for people with MS.

ELIGIBILITY:
Inclusion Criteria:

* Neurologist-confirmed diagnosis of primary progressive or relapsing and remitting MS per The 2017 Revision of the McDonald Criteria and the Magnetic Resonance Imaging in MS, or a healthy volunteer without a diagnosis of multiple sclerosis or any related neurological conditions
* Fluent in speaking and understanding English
* Subjects with multiple sclerosis have self-reported vestibular symptoms of dizziness, imbalance, and/or a history of at least two falls in the prior 12 months

Exclusion Criteria:

* Clinically isolated syndrome or radiologically isolated syndrome.
* Worsening MS symptoms during the prior 60 days
* Immunotherapy change in the prior 60 days
* Self-reported cognitive impairment that limits independence with basic and instrumental activities of daily living
* Systolic blood pressure > 180 mmHg and/or diastolic blood pressure > 90 mmHg at rest
* Static visual acuity with correction of worse than 1.0 logMAR
* Manifest ocular misalignment ≥ 5 diopters (e.g., tropia, lazy eye, strabismus}
* Convergence insufficiency
* Intra-nuclear ophthalmoplegia
* Vestibular Migraine
* Major orthopedic conditions that limit cervical spine range of motion or that alter walking
* Self-reported current or potential for pregnancy during enrollment
* Ongoing participation in vestibular rehabilitation for dizziness

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Composite VOR gain (cVOR gain) | Weeks 0,1,2,3,4,5,6, 7, and 18
  The team will conduct the video head impulse test (vHIT), a physiologic assay of vestibular semicircular canal pathway function. Angular vestibulo-ocular reflex gain will be calculated as eye velocity / head velocity during self-generated and/or passive high frequency head rotations which will be conducted in the yaw, pitch, roll, and/or semicircular canal planes.

SECONDARY OUTCOMES:
Best Corrected Dynamic Visual Acuity (During Head Movements) | Weeks 0,1, 4, 7, and 18
  The ability of participants to see clearly while their head is in motion (e.g., during self-generated head movements while seated, while walking at their preferred walking speed) will be assessed using commercially available hardware and custom software while the participant's head is moving.
Balance Evaluation Systems Test Total Score | Weeks 1, 4, 7, and 18
  The BEST will be instrumented using inertial measurement units (IMU) placed at the head, upper torso, pelvis, and both ankles. The BEST is a 36-item assessment of the body systems that contribute to balance and walking. Total scores range from 0 to 108 points
Gait Disorientation Test (GDT) Score | Weeks 1, 4, 7, and 18
  The GDT is a 2-item assessment of aspects of spatial navigation. Task 1 is to walk 20 feet with eyes open. Task 2 is to walk 20 feet with eyes closed. Both tasks are timed, and the GDT result is the time needed to walk with eyes closed minus the time needed to walk with eyes open.
Dizziness Handicap Inventory Total Score | Weeks 1, 4, 7, and 18
  The DHI be used to assess participants' perceived level of handicap due dizziness. This measure consists of 25 questions that are answered as "yes" = 4 points (dizziness is always a factor), "sometimes" = 2 points (dizziness is sometimes a factor), or "no" = 0 points (dizziness is never a factor) for a given situation or issue. The maximum total score on this measure is 100 points with higher scores indicating higher levels of perceived handicap.
Activities-specific Balance Confidence Scale Average Score | Weeks 1, 4, 7, and 18
  The ABCS consists of 16 questions for which the respondent answers how confident they feel in not becoming unsteady or falling in specific situations. Confidence is rated on a scale of 0% to 100% with 0% indicating "no confidence" and 100% indicating "complete confidence' in the ability to maintain balance. Average scores of ≥ 80% are associated with high levels of physical functioning in adults.
Oscillopsia Visual Analog Scale Score | Weeks 1, 4, 7, and 18
  Visual analog scales are commonly used in clinical practice and research. The investigator will measure the severity of oscillopsia (unstable vision during head movement) and sense of disequilibrium while the participant walks 20' on separate visual analog scales. The distance from the zero anchor to the respondent's marking will be measured without units but to the nearest tenth. The response for each scale will be transformed to a 100-point scale
Disequilibrium Visual Analog Scale Score | Weeks 1, 4, 7, and 18
  The investigator will measure the sense of disequilibrium while the participant walks 20' on separate visual analog scales. The distance from the zero anchor to the respondent's marking will be measured without units but to the nearest tenth.
  The response for the scale will be transformed to a 100-point scale.
Multiple Sclerosis Quality of Life - 54 (MSQOL-54) Total Score | Weeks 1, 4, 7, and 18
  The MSQOL-54 is a multidimensional measure that consists of questions related to general and MS-specific health-related quality of life. The MSQOL-54 was created by adding 18 items related to MS-specific issues, e.g., fatigue and cognitive function.
Global Perception of Effect Score | Weeks 1, 4, 7, and 18
  The investigator will assess perception of change retrospectively across the entire study period with ratings using an 11-point Likert scale with anchors of "very much better" and "very much worse" with a middle point labeled "no change" to assess the magnitude of change in symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Grove, PT, MS, DPT, PhD, Principal Investigator — Emory University
Locations (1):
- Emory Univeristy, Atlanta, Georgia, United States